CLINICAL TRIAL: NCT03840382
Title: Telemedicine for PrEP Throughout Mississippi
Acronym: Tele-PrEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Larry K. Brown, Director, Division of Child and Adolescent Psychiatry, Rhode Island Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 407618
Record Dates: First submitted 2019-01-28; First posted 2019-02-15 (Actual); Results first posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2023-11

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tele-PrEP Intervention (Experimental): The telemedicine intervention will allow participants to discuss HIV prevention and PrEP with PrEP specialists at an academic medical center via videoconference from their local community based organization (CBO). During the intervention, participants will gain information related to HIV and PrEP, view a video to improve motivation for engagement in PrEP related care, and receive resources to address barriers to care.
  Interventions: Behavioral: Tele-PrEP Intervention

INTERVENTIONS:
Behavioral: Tele-PrEP Intervention — Telemedicine conferences with PrEP-specialists

SUMMARY:
This study will develop and test a program to deliver PrEP care in underserved communities in Mississippi (MS) through telemedicine, distance-based, clinical care delivered in local community based organizations (CBOs). The intervention will be developed in collaboration with medical specialists at the University of Mississippi Medical Center (UMMC) and local CBO stakeholders (providers, administrators and patients). Approximately 75 individuals will be recruited from CBOs in MS. Participants will be able to receive PrEP counseling in the CBO and PrEP care via telemedicine from a PrEP specialist at UMMC. Participants will complete three assessments in the six months after enrolling. Our study will provide a wealth of information about PrEP-related outcomes and HIV testing among MS residents living in underserved communities. If successful, this program will be able to be disseminated to other CBOs in the South.

DETAILED DESCRIPTION:
Uptake of PrEP in the southern United States has been slow, especially in areas distant from academic medical centers that provide PrEP care. Despite underserved populations in the South having alarmingly high rates of HIV, a large percentage of at-risk individuals are not engaged in PrEP care due to limited access to academic medical centers. Mississippi (MS), the site of this proposed project, has the seventh highest incidence of HIV of any state and CBOs that provide HIV/STI testing outside of urban areas report that very few of their at-risk individuals use PrEP. Unfortunately, physicians outside of academic centers are often reluctant to prescribe PrEP because they lack the expertise, training, and the support necessary to provide comprehensive HIV prevention care. Those are at-risk do not seek PrEP from academic centers because of stigma, travel burdens, and financial concerns. To overcome these barriers, this project will develop and pilot test a program to deliver PrEP care in underserved remote communities in MS through telemedicine clinical care delivered in local CBOs. Telemedicine will allow specialists to provide care at a distance and while simultaneously enhancing the capacity of local CBOs to provide quality HIV testing and counseling, PrEP treatment, and linkage to HIV care if needed. It will allow patients to receive the highest level of medical care from trusted CBOs within their local communities. It will also enhance the CBO's mission by allowing it to provide a new, high-quality medical service.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Presented at a collaborating CBO for HIV testing during trial months
* PrEP eligible based on HIV Risk Checklist
* Able to read and speak English
* Able to give meaningful consent as determined by research staff
* No known HIV infection

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry K Brown, MD, Principal Investigator — Rhode Island Hospital; James B Brock, MD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tele-PrEP Intervention
Started | 74
Completed | 63
Not Completed | 11
Not completed — Lost to Follow-up | 11

BASELINE CHARACTERISTICS:
Population: Participants who completed the baseline assessment.
Arm/Group | Tele-PrEP Intervention
Number analyzed (Participants) | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.3 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 60
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 51
  White | 9
  More than one race | 1
  Unknown or Not Reported | 1
PrEP knowledge [Mean (Standard Deviation); unit: score on a scale] — 5-item questionnaire to assess knowledge (true/false/don't know) based on facts from the CDC and the San Francisco AIDS Foundation websites concerning PrEP.
  The score of this measure ranges from 0 to 5, with 5 indicating higher levels of PrEP knowledge.
  score on a scale | 2.63 (1.72)
Motivational readiness for PrEP and PrEP-related care [Mean (Standard Deviation); unit: score on a scale] — This measure was a subscale adapted from The LifeWindows Information Motivation Behavioral Skills ART Adherence Questionnaire (LW-IMB-AAQ), 2006. The motivational readiness to engage in PrEP care subscale consisted of eight items with 4-point Likert responses. The possible score range for this subscale is 8 to 32, with higher scores indicating higher motivation to engage in PrEP care. Population: Only those who completed 80% of the scale or more are included in the analyses. This explains why the number analyzed for this measure is lower than the overall number of baseline participants.
  score on a scale
    number analyzed (Participants) | 61
    (all) | 25.07 (4.37)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Attended One or More PrEP Telemedicine Appointments at 3 Months Post-intervention (Electronic Medical Record Extraction)
Description: Number of participants who attended one or more PrEP telemedicine appointments with a UMMC PrEP specialist, in the past 3 months, extracted from patient's electronic medical record at 3 months post-intervention.
Time Frame: Assessed at 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Tele-PrEP Intervention
Number analyzed (Participants) | 63
Participants | 8

2. Primary Outcome: Number of Participants Who Attended One or More PrEP Telemedicine Appointments at 6 Months Post-intervention (Electronic Medical Record Extraction)
Description: Number of participants who attended one or more PrEP telemedicine appointments with a UMMC PrEP specialist, in the past 3 months, extracted from patient's electronic medical record at 6 months post-intervention.
Time Frame: Assessed at 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Tele-PrEP Intervention
Number analyzed (Participants) | 63
Participants | 2

3. Primary Outcome: Number of Participants Who Received a PrEP Medication Prescription at 3 Months (Electronic Medical Record Extraction)
Description: Number of participants who received a PrEP medication prescription in past 3 months, extracted from patient's electronic medical record at 3-month follow-up.
Time Frame: Assessed at 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Tele-PrEP Intervention
Number analyzed (Participants) | 63
Participants | 22

4. Primary Outcome: Number of Participants Who Received a PrEP Medication Prescription at 6 Months (Electronic Medical Record Extraction)
Description: Number of participants who received a PrEP medication prescription in past 3 months, extracted from patient's electronic medical record at 6-month follow-up.
Time Frame: Assessed at 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Tele-PrEP Intervention
Number analyzed (Participants) | 63
Participants | 17

5. Primary Outcome: Adherence to PrEP (Self-report)
Description: Self-reported number of days a PrEP dose was missed in the past 30 days. Ranging from 0 to 30.
Time Frame: Assessed at 3 months and 6 months
Population: Only participants who self-reported current PrEP use were included in these analyses.
Measure: Mean (Standard Deviation); unit: missed PrEP doses
Arm/Group | Tele-PrEP Intervention
Number analyzed (Participants) | 28
missed PrEP doses
  Missed Doses at 3-Months | 2.07 (3.03)
  Missed Doses at 6-Months | 18.75 (13.50)

6. Primary Outcome: Number of Participants With 0-2 PrEP Refills at 3 Months (Electronic Medical Record )
Description: Number of participants with 0-2 PrEP medication refills in past 3 months (extracted from electronic medical record at 3-month follow-up).
Time Frame: Assessed at 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Tele-PrEP Intervention
Number analyzed (Participants) | 63
Participants
  0 Refills | 43
  1 Refill | 11
  2 Refills | 9

7. Primary Outcome: Number of Participants With 0-2 PrEP Refills at 6 Months (Electronic Medical Record)
Description: Number of Participants With 0-2 PrEP Refills in past 3 months (extracted from electronic medical record at 6-month follow-up).
Time Frame: Assessed at 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Tele-PrEP Intervention
Number analyzed (Participants) | 63
Participants
  0 Refills | 46
  1 Refill | 12
  2 Refills | 5

8. Secondary Outcome: PrEP Knowledge
Description: This 5-item measure was used to assess knowledge (true/false/don't know) based on facts from the CDC and the San Francisco AIDS Foundation websites concerning PrEP.
  Scores for the measure could range from 0 to 5 with higher scores indicating greater PrEP knowledge.
Time Frame: Assessed at 3 months and 6 months
Population: Only those who completed 80% of the scale or more are included in the analyses. This is why only 57 and 54 participants were included in the 3-month and 6-month analysis, respectively.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tele-PrEP Intervention
Number analyzed (Participants) | 63
score on a scale
  Score at 3-months: number analyzed (Participants) | 57
  Score at 3-months | 2.89 (1.84)
  Score at 6-months: number analyzed (Participants) | 54
  Score at 6-months | 2.93 (1.64)

9. Secondary Outcome: Motivational Readiness for PrEP and PrEP-related Care
Description: This measure was a subscale adapted from The LifeWindows Information Motivation Behavioral Skills ART Adherence Questionnaire (LW-IMB-AAQ), 2006. The motivational readiness to engage in PrEP care subscale consisted of eight items with 4-point Likert responses. The possible score range for this subscale is 8 to 32, with higher scores indicating higher motivation to engage in PrEP care.
Time Frame: Assessed at 3 months and 6 months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tele-PrEP Intervention
Number analyzed (Participants) | 63
score on a scale
  Score at 3-Months: number analyzed (Participants) | 57
  Score at 3-Months | 25.95 (4.69)
  Score at 6-Months: number analyzed (Participants) | 54
  Score at 6-Months | 26.50 (4.11)

10. Secondary Outcome: Patient Acceptability Score Regarding the Use of Telemedicine for PrEP Care (CSQ-8)
Description: Patients' perspective on the acceptability of using telemedicine for PrEP care was assessed with a modified version of the Client Satisfaction Questionnaire (CSQ-8). This measure was only given to participants who attended a PrEP-related telemedicine appointment. Scores for this measure could range from 2 to 8, with higher scores indicating greater satisfaction.
Time Frame: Assessed at 3 months and 6 months
Population: Only those who attended a telemedicine for PrEP appointment and completed this measure on the survey were included in the analyses. By 3-month follow-up, 11 of 63 participants used telemedicine for PrEP care. By 6-month follow-up, 1 additional participant used telemedicine for PrEP care. This explains why the overall number of participants analyzed for this measure was 12, as opposed to 63.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tele-PrEP Intervention
Number analyzed (Participants) | 12
score on a scale
  Score at 3-Months: number analyzed (Participants) | 11
  Score at 3-Months | 7.27 (1.27)
  Score at 6-Months | 7.50 (1.00)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the 6 month study duration.
Arm/Group | Tele-PrEP Intervention
All-Cause Mortality (participants affected / at risk) | 0/63
Serious Adverse Events (participants affected / at risk) | 0/63
Other Adverse Events (participants affected / at risk) | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-12): https://cdn.clinicaltrials.gov/large-docs/82/NCT03840382/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-27): https://cdn.clinicaltrials.gov/large-docs/82/NCT03840382/ICF_001.pdf